CLINICAL TRIAL: NCT02321865
Title: Dose Adjustment Study of NPC-02 in Patients With Zinc Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-02-5
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2015-07

CONDITIONS: Zinc Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NPC-02 (Experimental)
  Interventions: Drug: NPC-02

INTERVENTIONS:
Drug: NPC-02

SUMMARY:
The objective of this study is to check the dose control method of NPC-02 and the holding effect for the target serum zinc concentration in patients with zinc deficiency.

ELIGIBILITY:
Inclusion Criteria:

* The serum zinc concentrations are under the nomal level before registration
* Able to taking a tablet

Exclusion Criteria:

1. Heavy hepatitis
2. Malignant tumor
3. Severe heart disease, hematological disorder, kidney disease and pancreatic disease, etc.
4. The serum albumin under 2.8 g/dL
5. Patient of allergy and hyperesthesia to zinc containing medicine manufacturing (including supplement)
6. Patient who was taking a medicine including the zinc (including supplement) within 12 weeks before registration
7. Pregnant, suspected pregnant, lactating, patients who wish to have a child
8. Patient who participated in other clinical trials within 12 weeks before registration
9. Unsuitable as a target of this clinical trial judged by doctor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11-24 (Actual)

PRIMARY OUTCOMES:
The ratio of the patients who could maintain target serum zinc concentration | approx. 12-24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka, Japan

REFERENCES:
- [Derived] Katayama K, Hosui A, Sakai Y, Itou M, Matsuzaki Y, Takamori Y, Hosho K, Tsuru T, Takikawa Y, Michitaka K, Ogawa E, Miyoshi Y, Ito T, Ida S, Hamada I, Miyoshi K, Kodama H, Takehara T. Effects of Zinc Acetate on Serum Zinc Concentrations in Chronic Liver Diseases: a Multicenter, Double-Blind, Randomized, Placebo-Controlled Trial and a Dose Adjustment Trial. Biol Trace Elem Res. 2020 May;195(1):71-81. doi: 10.1007/s12011-019-01851-y. Epub 2019 Aug 7. PMID 31392541